CLINICAL TRIAL: NCT00862225
Title: Randomized, Double-blind Prospective Clinical Study to Examine the Mechanism of Action of IG-RD-001 (Ze-339) Compared to Desloratadine and Placebo in Patients With Seasonal Allergic Rhinitis Who Are Sensitized to Grasses
Brief Title: MOA Study of Ze 339 in Seasonal Allergic Rhinitis
Acronym: PETRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Max Zeller Soehne AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PETRA_IG-RD-001 (Ze339); EudraCT-Number: 2007-006090-89
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: rhinomanometry; mode of action; grass pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Ze 339

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Desloratadin
- 3 (Experimental)
  Interventions: Drug: IG-RD-001 / Ze 339

INTERVENTIONS:
Drug: Placebo — Following a 3-way crossover treatment design (IG-RD-001 (Ze 339), desloratadine, placebo), a controlled, unilateral, nasal allergen provocation (grasses) will be carried out on 18 study participants. The time-dependent development of the nasal obstruction, measured via rhinomanometry before and after the allergen provocation, will be the effect parameter.
  Arms: 1
Drug: Desloratadin — Following a 3-way crossover treatment design (IG-RD-001 (Ze 339), desloratadine, placebo), a controlled, unilateral, nasal allergen provocation (grasses) will be carried out on 18 study participants. The time-dependent development of the nasal obstruction, measured via rhinomanometry before and after the allergen provocation, will be the effect parameter.
  Arms: 2
Drug: IG-RD-001 / Ze 339 — Following a 3-way crossover treatment design (IG-RD-001 (Ze 339), desloratadine, placebo), a controlled, unilateral, nasal allergen provocation (grasses) will be carried out on 18 study participants. The time-dependent development of the nasal obstruction, measured via rhinomanometry before and after the allergen provocation, will be the effect parameter.
  Arms: 3

SUMMARY:
Randomised, double-blind and prospective clinical study to examine the mechanism of action of the Petasites hybridus leaf extract IG-RD-001 (Ze-339, petasol butenoate complex) compared to desloratadine and placebo in patients with seasonal allergic rhinitis of all degrees of severity (provoked by grasses). The treatment arm with desloratadine is an established standard treatment and is intended to ensure the comparative methodology of the study.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis since at least 2 years
* Age: = > 18 years
* Consent in accordance with the AMG (=German Drug Law)
* Positive skin test, skin prick test or positive RAST for grasses The skin prick test is positive if the wheal is >= 3 mm greater than control; a skin test is positive if the wheal is >= 7 mm greater than control
* Women of childbearing potential have to use a highly effective method of birth control (according CPMP/ICH/286/95 Note 3) during the duration of the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.

Exclusion Criteria:

* Past or current psychological disease or disorder which can impair the study participant's ability to understand the study requirements, t take part in the study or give consent after briefing
* Past or current alcohol or medication dependency or abuse
* Bronchial asthma (FEV < 80 %)
* Glaucoma, cataract or ocular herpes simplex
* Clinically relevant deviations from normal laboratory parameters (if known)
* Antihistamines with a long-term effect
* Malignant diseases, including in the patient's case history
* Parasites
* Study participants who are taking part in another study or took an investigational product during the last 4 weeks before the start of treatment
* Progressive systemic diseases such as tuberculosis, leukoses, collagenoses, multiple sclerosis, Aids, HIV infection and other autoimmune diseases
* Other types of rhinitis with different causes, acute or chronic sinusitis
* Pregnancy or lactation
* Serious internal diseases, e.g. serious decompensated diseases of the heart, liver, kidneys or diabetes mellitus
* Patients with rarely occurring hereditary problems galactose-intolerance, Lapp-lactase-deficiency or glucose-galactose-malabsorption
* Pre-existing liver damage
* The use of non-steroidal antirheumatic agents (NSAR)
* Hypersensitivity towards one of the ingredients in the investigational product
* Not adhering to the following periods of abstention before the nasal provocation test: 3 days for DNCG, nedocromil, nasal and oral antihistamines, and tricyclic psychotropic drugs, 1 months systemic treatment with glucocorticoids, 14 days for nasal and topical corticosteroids, 1 week for antihistamines, and 1 day for α-adrenergic drugs. The use of ACE inhibitors or ß-blockers
* Previous organ transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The time-dependent development of the nasal obstruction, measured via rhinomanometry before and after the allergen provocation, will be the effect parameter. | 0-24 hours post nasal provocation test

SECONDARY OUTCOMES:
Clinical symptom score (rhinorrhoea, nasal congestion, nasal itching and sneezing), assessment by the investigator (nasal secretion, irritation, occurrence of systemic symptoms), mediators in the serum, nasal secretion, nasal curettage and biopsy | 0-24h post nasal provocation test

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Otorhinolaryngology and Head and Neck Surgery, Düsseldorf, Germany

REFERENCES:
- See also: Link to publication in PubMed — http://www.ncbi.nlm.nih.gov/pubmed/21489609